CLINICAL TRIAL: NCT03108638
Title: Supporting Sustainable Positive Interactions in the Child Welfare System: The R3 Supervisor Strategy
Acronym: R3
Status: Completed | Type: Observational
Sponsor: Oregon Social Learning Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Other Study IDs: R01DA040416 (NIH); R01DA040416 (NIH)
Record Dates: First submitted 2016-06-14; First posted 2017-04-11 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-11

CONDITIONS: Behavioral
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- R3 Supervisor Strategy Region 1: First cohort to be trained and monitored with remote coaching in the R3 model
  Interventions: Behavioral: R3 Supervisor Implementation Strategy
- R3 Supervisor Strategy Region 2: Second cohort to be trained and monitored with remote coaching in the R3 model
  Interventions: Behavioral: R3 Supervisor Implementation Strategy
- R3 Supervisor Strategy Region 3: Third cohort to be trained and monitored with remote coaching in the R3 model
  Interventions: Behavioral: R3 Supervisor Implementation Strategy
- R3 Supervisor Strategy Region 4: Fourth cohort to be trained and monitored with remote coaching in the R3 model
  Interventions: Behavioral: R3 Supervisor Implementation Strategy

INTERVENTIONS:
Behavioral: R3 Supervisor Implementation Strategy — Supervisors will be trained to provide supervision to their caseworkers using R3 principles and strategies. Monthly monitoring and remote coaching will be provided.
  Other Names: R3

SUMMARY:
Opportunities to implement and evaluate system-wide change are rare. This observational, Hybrid II study leverages a real-world, system-initiated roll-out of R3, a supervisor-targeted implementation strategy aimed at infusing the use of evidence-based principles across multiple levels of the workforce within a public child welfare system. This project aims to study the effectiveness of R3 in impacting organizational inner-context variables and subsequent positive outcomes for one of the nation's most costly and vulnerable populations-families involved in the child welfare system.

DETAILED DESCRIPTION:
Large knowledge gaps remain regarding strategies to promote change in public child welfare systems (CWS), yet opportunities to evaluate strategies to create system-wide change and the resulting public health impact are rare. The CWS in the United States is populated with vulnerable children and families at high risk for negative outcomes, including substance use, risky sexual behavior, delinquency, incarceration, homelessness, and early mortality. This proposal addresses the National Institute of Health (NIH) priority to understand methods for "scale-up and sustainability of evidence-based interventions." Leveraging a real-world, federally funded, system-initiated effort to infuse the use of evidence-based principles throughout the multi-levels of the Tennessee CWS workforce, this study will evaluate the effectiveness of a supervisor-targeted implementation strategy in creating organizational change and subsequent positive family outcomes. The R3 Supervisor Strategy was developed to modify the way that the CWS workforce supports families toward completing their treatment plans, by utilizing evidence-based behavioral principles found in previous intervention trials to improve system-level outcomes, including child permanency, stability, and well-being. The R3 strategy provides training, consultation, and fidelity-monitoring to supervisors, who are centrally positioned in the system between caseworkers (who have daily interactions with CWS-involved families) and leadership (who make decisions that affect the organization in which families receive services). The three Rs include reinforcement of (1) effort, (2) relationships and roles, and (3) small steps toward goal achievement. R3 is founded on social learning theory; these reinforcement targets are encouraged in interactions between supervisors and their supervisee- caseworkers and between caseworkers and the families they serve. Utilizing a variation of a dynamic wait-listed design, four Tennessee CWS regions (serving over 12,000 children annually) that have been awarded a federal Title-IV-E Waiver and have opted to adopt R3 as part of their waiver plan will be observed. The CWS workforce (n = 85 regional administrators, 50 supervisors, and 220 caseworkers) will be recruited to participate in a Hybrid Type II trial of the effectiveness of R3 in achieving organizational and subsequent positive system-level, client-level outcomes. This project will examine the potential of R3 to influence supervisor interactions with caseworkers and subsequent family outcomes (Aim 1); the impact of R3 on organizational characteristics known to impact staff retention and the successful adoption of innovations such as climate, leadership, readiness, and citizenship (Aim 2); and the potential for maintaining fidelity standards to the R3 strategy as consultation and coaching are fully transferred to the system (Aim3). This project will inform the potential for R3 to effectively infuse evidence-based principles into the daily interactions of those involved in the CWS, and to narrow the gap for achieving outcomes for one of the nations most costly and vulnerable populations-families involved in the child welfare system.

ELIGIBILITY:
Inclusion Criteria:

* Child Welfare Workforce in the state of Tennessee

Exclusion Criteria:

* Contract Workers

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population being studied is the child welfare workforce including supervisors and their staff
Sampling Method: Non-Probability Sample
Enrollment: 531 (Actual)
Dates: Start 2015-09-15 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Examination of child welfare supervisor ratings using the Fidelity of R3 Implementation for Supervisors (FRI_S) standardized measurement. | Monthly for 3 years from baseline to 36 months
  The Fidelity of R3 Implementation for Supervisors (FRI_S) measure will be used to rate supervisors' monthly delivery of the R3 model with fidelity over time, from baseline to 36 months.

SECONDARY OUTCOMES:
Organizational Climate, Leadership, Readiness, Attitudes toward Evidence-Based Practice: | Once a year for 3 years
  Organizational health and factors known to be related to successful adoption of new practices will be collected from child welfare staff members annually for 3 years.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Saldana, PhD, Principal Investigator — OSLC

IPD SHARING:
Plan to Share IPD: No